CLINICAL TRIAL: NCT01253850
Title: Improving Antiretroviral Medication Adherence Among HIV-infected Youth: Phase I
Status: Completed | Type: Observational
Sponsor: Fenway Community Health (Other)
Collaborators: Massachusetts General Hospital (Other); Boston Children's Hospital (Other); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Matthew Mimiaga, Research Scientist, Fenway Community Health
Other Study IDs: CFAR Adherence HIV Youth:1
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: HIV Infection
Keywords: hiv; antiretroviral; adherence; adolescent
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
HIV is increasing among adolescents and young adults in the US. Antiretroviral medications, when taken correctly (≥90% of prescribed doses taken), can vastly improve life expectancy. However, adherence among HIV-infected young people is suboptimal, and few interventions are available to help adolescents adhere to treatment.

The first phase of the study is an intervention development phase, which includes conducting interviews with 40 HIV-infected youth for input on the adaptation of the approach. The information obtained from the qualitative interviews is used to adapt the Life-Steps intervention (designed by our group for HIV-infected adults) to be responsive to the needs of HIV-infected adolescents, with acceptability of topics and content, and feasibility of intervention delivery to be tested in an open pilot trial.

DETAILED DESCRIPTION:
This phase of the protocol focuses on setting up the infrastructure necessary for conducting the study, including hiring and training activities with study staff. This time will be spent conducting interviews and using these data to inform the development of the intervention protocol and adaptation of all Life-Steps intervention materials, including study assessment instruments, for HIV-infected youth.

The interview is a one-time event and will last for 1.5-2 hours. It has two components: a quantitative assessment and a qualitative discussion. After all participants have completed the informed consent and assent (if under the age of 18) processes, the research staff will administer a brief quantitative assessment that will ask questions related to demographics, medication adherence, sexual risk, substance use, and psychosocial condition. The second part of the interview will be an open discussion. The interviews will be conducted by a trained member of the research staff. The interviews will be informed by a pre-determined qualitative topic guide.

ELIGIBILITY:
Phase I

Inclusion Criteria:

* Age 13 to 24 years
* HIV-infected and aware of HIV-infection status
* Currently taking antiretroviral therapy, has been prescribed antiretroviral therapy in the past 6 months, or a medical provider has recommended antiretroviral medications within the last 6 months
* Willing and able to provide informed consent or assent (if under the age of 18)

Exclusion Criteria:

* Not willing or able to provide informed consent or assent (if under the age of 18)
* Is dealing with a severe mental illness requiring immediate treatment (e.g. active psychotic episode) or a mental illness that would limit a participant's ability to engage with study protocol (e.g. dementia)
* Has severe cognitive limitations that would limit a participant's ability to comprehend the informed consent or assent.

Phase II

Inclusion Criteria:

* Age 13-24 years
* HIV-infected and aware of HIV-infection status
* Currently taking antiretroviral therapy
* Self-reported difficulties adhering to HIV medications in the past 3 months
* Self-identify as heterosexual or LGB
* Willing and able to provide informed consent/consent of parent/guardian if under the age of 18

Exclusion Criteria:

* Not willing or able to provide informed consent or assent (if under the age of 18)
* Is dealing with a severe mental illness requiring immediate treatment (e.g. active psychotic episode) or a mental illness that would limit a participant's ability to engage with study protocol (e.g. dementia)
* Has severe cognitive limitations that would limit a participant's ability to comprehend the informed consent or assent.

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: HIV-infected youth between the ages of 13 and 24
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2010-08; Primary Completion 2011-07 (Actual); Study Completion 2013-03-06 (Actual)

PRIMARY OUTCOMES:
perceived barriers and facilitators to adherence | One-time qualitative interview
  We will code the qualitative interview data for key themes that emerge with respect to adherence and intervention needs. The information obtained from the qualitative interviews is used to adapt the Life-Steps intervention (designed by our group for HIV-infected adults) to be responsive to the needs of HIV-infected adolescents, with acceptability of topics and content, and feasibility of intervention delivery to be tested in an open pilot trial.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Mimiaga, ScD MPH, Principal Investigator — Fenway Health and Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - Fenway Community Health, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No